CLINICAL TRIAL: NCT05947110
Title: How Effective is the Plyometric-based Hydro-kinesio Therapy for Pain, Muscle Strength, Postural Control, and Functional Performance in Children With Hemophilic Knee Arthropathy?
Brief Title: Plyometric-Based Hydro-Kinesio Therapy in Children With Hemophilic Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0033
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Haemophilic Arthropathy of Knee

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyo-HKT group (Experimental): Participants in this group received the Plyo-HKT program
  Interventions: Other: Plyometric-based hydro-kinesio therapy
- Control group (Active Comparator): Participants in this group received the standard exercise program.
  Interventions: Other: Standard exercise therapy

INTERVENTIONS:
Other: Plyometric-based hydro-kinesio therapy — The plyometric-based hydro-kinesio therapy was conducted for 45 minutes, twice weekly, for 8 successive weeks. The training was geared toward the lower body and was conducted under the close supervision of a licensed pediatric physical therapist in accordance with the safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association.
  Arms: Plyo-HKT group
Other: Standard exercise therapy — The program encompassed the standard exercises for patients with JIA (aerobic, weight-bearing, proprioceptive, flexibility, and strengthening exercises). The training was conducted for 45 minutes, two times a week for 8 successive weeks.
  Arms: Control group

SUMMARY:
This study was designed to assess the effect of an 8-week plyometric-based hydro-kinesio therapy (Plyo-HKT) on pain, muscle strength, postural control, and functional performance in a convenience sample of children with hemophilic knee arthropathy (HKA). Forty-eight patients with HKA were randomly allocated to the Plyo-HKT group (n = 24, received the plyometric-based hydro-kinesio therapy program, twice/week, over 8 weeks) or the control group (n = 24, received standard exercise program). Both groups were assessed for pain, muscle strength, postural control, and functional performance pre and post-treatment.

DETAILED DESCRIPTION:
Forty-eight boys with moderate hemophilia-A were recruited from the hematology clinics of three large referral hospitals in Riyadh, Saudi Arabia. The study included patients who were 8-16 years old, had factor VIII replacement prophylaxis, were clinically-stable cases, had unilateral knee hemarthrosis, had grade II or III knee arthropathy, had muscle strength of grade three, and if they were able to walk independently. Patients who had enduring disabling pain, fixed deformities, a history of musculoskeletal surgery, visual and/or vestibular deficits, or bleeding episodes within two weeks before enrollment were excluded.

Outcome measures

Pain: Pain during rest and/or movement was assessed using the Numerical Pain Rating Scale.

Muscle strength: The peak concentric torque of the quadriceps and hamstring muscles was measured through an Isokinetic Dynamometer.

Postural control: The directional dynamic limit of stability (forward, backward, affected, and non-affected) and overall limit of stability were assessed using the Biodex balance system.

Functional performance: The extent of functional capacity was assessed through the functional independence score in hemophilia and the six-minute walk test.

Interventions

The Plyo-HKT group received the Plyo-HKT program, 45 minutes per session, two times a week for 8 consecutive weeks, in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The Plyo-HKT program consisted of ten unilateral and bilateral lower limb plyometrics in the form of hopping/bounding/jumping activities conducted in a water medium. The Plyo-HKT included a warm-up for 10 minutes and a cool-down for 5 minutes. The control group received the standard exercise program, 45 minutes per session, two times a week for 8 consecutive weeks. The program consisted of flexibility exercise, strength training, weight-bearing, proprioceptive training, and free treadmill walking or cycle ergometry.

ELIGIBILITY:
Inclusion Criteria:

* Eight and 16 years.
* Had factor VIII replacement prophylaxis.
* Clinically-stable.
* Unilateral knee involvement.
* Knee arthropathy of grade II or III per the Arnold-Hilgartner radiographic classification.
* Muscle strength of grade 3 in lower limb muscles.
* Use of no pain medication for one month prior to enrollment.
* Walking independently.

Exclusion Criteria:

* Enduring disabling pain
* Fixed deformities.
* History of musculoskeletal surgery.
* Visual or vestibular deficits.
* Engagement in regular exercises.
* Bleeding episodes within two weeks prior to enrolment.

Ages: 8 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 2 months
  Participants reported how much they feel pain during rest and/or movement on the 0-10 Numerical Pain Rating Scale, where 0 represents "no pain" and 10 indicates the "worst possible pain".
Muscle strength | 2 months
  Indicated by the peak concentric torque of the quadriceps and hamstring muscles (Nm). It was measured using an Isokinetic Dynamometer.
Postural control | 2 months
  The capacity to control and move the center of gravity in various directions across the base of support was assessed utilizing the Biodex balance system. Values are expressed as accuracy % and higher scores mean better balance capability.

SECONDARY OUTCOMES:
Functional independence | 2 months
  The functional independence was assessed using the Functional Independence Score in Hemophilia. The test includes an assessment of eight activities, divided into three categories (selfcare, transfer, and mobility). Each activity is rated on a 1-4 scale, where 1 indicates that participant was unable to execute the action or requires full support and 4 indicates being able to do the task without any difficulties. The maximum score is 32, which denotes the highest degree of independence.
Six-minute walk test | 2 months
  The six-minute walk test measured the walking distance that children were able to cover across a 30-m walkway with a self-determined walking pace over six minutes. A longer distance indicates a better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia